CLINICAL TRIAL: NCT03031548
Title: Intraoperative Point-of Care Ultrasound for Identification of Endotracheal Tube Position in the Pediatric Population
Brief Title: Intra-op POCUS for Identification of Endotracheal Tube Position in the Pediatric Population
Acronym: POCUS
Status: Completed | Type: Observational
Sponsor: Loma Linda University (Other)
Responsible Party: Principal Investigator, Elizabeth Ghazal, Principal Investigator, Loma Linda University
Other Study IDs: 5160372
Record Dates: First submitted 2017-01-09; First posted 2017-01-25 (Estimated); Last update posted 2021-03-15 (Actual); Status verified 2021-03

CONDITIONS: Endotracheal Tube Wrongly Placed During Anesthetic Procedure

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (1):
- ultrasound exam: Child undergoing procedure in CVL requiring ETT and CXR as standard of care - received point-of-care ultrasound exam as part of the study
  Interventions: Device: Point-of-care ultrasound exam; Radiation: Reposition ETT

INTERVENTIONS:
Device: Point-of-care ultrasound exam — No intervention
  Other Names: POC ultrasound
Radiation: Reposition ETT — ETT will be repositioned based on CXR by fluoroscopy

SUMMARY:
Chest X-ray and/or fluoroscopy is not routinely used in the OR to confirm endotracheal tube (ETT) placement by anesthesiologists. Multiple studies have shown that ~19% of all intubations result in inappropriate ETT placement. An adult study has shown that ultrasound point-of-care is superior to auscultation in determining the location of ETT. This study aims to determine if point-of-care is useful in determining ETT position in children.

DETAILED DESCRIPTION:
Patients scheduled to have a procedure in the cardiovascular laboratory where fluoroscopy is routinely used will also undergo a point-of-care ultrasound exam to determine endotracheal tube position. An anesthesiologist will perform the ultrasound exam.

ELIGIBILITY:
Inclusion Criteria:

1. children birth to 10 years of age;
2. undergoing cardiac catheterization in the cath lab;
3. general anesthesia with an endotracheal tube;
4. subjects will also receive a chest x-ray as standard of care

Exclusion Criteria:

1. children ages birth to 10 years undergoing cardiac catheterization under GA without an endotracheal tube;
2. emergency procedures;
3. known airway anomalies;
4. children who are non-English and non-Spanish speaking -

Ages: 1 Minute to 10 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child
Study Population: Children who require general anesthesia and endotracheal intubation for procedures in the cardiovascular laboratory
Sampling Method: Non-Probability Sample
Enrollment: 50 (Actual)
Dates: Start 2017-02-16 (Actual); Primary Completion 2018-06-30 (Actual); Study Completion 2018-06-30 (Actual)

PRIMARY OUTCOMES:
Endotracheal Tube Position | through study completion, an average of 1 year
  The primary outcome marker for this study was the correlation between the weighted POCUS measurement of TT location and the weighted fluoroscopy measurement of TT location

CONTACTS AND LOCATIONS:
Overall Officials: Elizabeth Ghazal, MD, Principal Investigator — Loma Linda University Health
Locations (2):
- United States (2):
  - Loma Linda University Health, Loma Linda, California
  - Loma Linda University Department of Anesthesiology, Loma Linda, California

IPD SHARING:
Plan to Share IPD: No